CLINICAL TRIAL: NCT06950801
Title: Comparing the Effects of Indoor vs. Outdoor Horticultural Therapy on College Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ye Zhiyin (Other)
Responsible Party: Sponsor-Investigator, Ye Zhiyin, Teaching assistant, Central University of Finance and Economics, China
Organization: Central University of Finance and Economics, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cufe03
Record Dates: First submitted 2025-03-04; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- outdoor-horticultural (Experimental): The participants in outdoor horticultural therapy engaged in weekly horticultural therapy activities outdoors for a total duration of eight weeks.
  Interventions: Behavioral: outdoor-horticultural therapy
- indoor-Horticultural (Experimental): The participants in indoor horticultural therapy engaged in therapeutic gardening activities indoors once a week for a total duration of eight weeks.
  Interventions: Behavioral: indoor-Horticultural Therapy group
- General Psychological Group (Placebo Comparator): Participants in the control group attended weekly psychological group sessions (without horticultural elements) for a total duration of eight weeks.
  Interventions: Behavioral: General Psychological Group Counselling Team
- Blank control group (No Intervention): These participants did not engage in any psychological activities; they only regularly took part in questionnaire completion.

INTERVENTIONS:
Behavioral: outdoor-horticultural therapy — Students are randomly assigned to the Outdoor Horticultural Therapy group, where they will receive outdoor horticultural therapy for eight weeks
  Arms: outdoor-horticultural
Behavioral: indoor-Horticultural Therapy group — Students are randomly assigned to the indoor horticultural therapy group, where they will receive indoor horticultural therapy for 8 weeks
  Arms: indoor-Horticultural
Behavioral: General Psychological Group Counselling Team — Students were randomly assigned to general group groups to participate in an 8-week mental health group activity
  Arms: General Psychological Group

SUMMARY:
This study used a randomised controlled trial to investigate the effects of different forms of horticultural group interventions on college students' depression, anxiety and subjective well-being, and the internal mechanisms of the effects.

Participants are required to complete the following tasks:

Attend one indoor/outdoor group gardening activity per week, lasting 2 hours each session, for a total of 8 weeks.

Complete psychological scale assessments at five time points: before the activity begins, at 4 weeks after the start, upon completion of the activity, and at 1 week and 2 weeks after completion.

ELIGIBILITY:
Inclusion Criteria:

- University students

Exclusion Criteria:

* Diagnosed with a mental disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Depression | From enrollment to 2 weeks after the completion of the 8-week treatment Edit Copy Outcome
  The Patient Health Questionnaire 9-item (PHQ-9): This scale consists of 9 items, each rated on a 4-point Likert scale, with higher scores indicating more severe depressive symptoms in the subject.
Anxiety | From enrollment to 2 weeks after the completion of the 8-week treatment
  Generalized Anxiety Disorder 7-item Scale (GAD-7): This scale consists of 7 items, each rated on a 4-point Likert scale, with higher scores indicating more severe anxiety symptoms in the subjects.
Positive And Negative Affective | From enrollment to 2 weeks after the completion of the 8-week treatment
  Positive and Negative Affect Schedule (PANAS): This scale consists of 20 items, including 10 positive affect items and 10 negative affect items, with each item rated on a Likert five-point scale. Higher scores on the positive affect items indicate higher levels of positive affect in the participants, while higher scores on the negative affect items indicate higher levels of negative affect in the participants.
Life satisfaction | From enrollment to 2 weeks after the completion of the 8-week treatment
  The Satisfaction With Life Scale (SWLS): This scale consists of 5 items, each rated on a 7-point Likert scale, with higher scores indicating greater life satisfaction among participants.

SECONDARY OUTCOMES:
Resilience | From enrollment to 2 weeks after the completion of the 8-week treatment
  The Connor-Davidson Resilience Scale (CD-RISC): The scale consists of 25 items divided into three dimensions-tenacity, self-reliance, and optimism. Each item is rated on a Likert five-point scale. Higher scores indicate greater psychological resilience in the subjects.
Loneliness | From enrollment to 2 weeks after the completion of the 8-week treatment
  UCLA Loneliness Scale: This scale consists of 8 items, each rated on a 5-point Likert scale, with higher scores indicating stronger feelings of loneliness in the subjects.
Sense of control | From enrollment to 2 weeks after the completion of the 8-week treatment
  Sense of Mastery Scale (SMS): This scale consists of 7 items, each using a 5-point Likert scale, with higher scores indicating a stronger sense of mastery in the subjects.
Avoidance | From enrollment to 2 weeks after the completion of the 8-week treatment
  The Brief Experiential Avoidance Questionnaire (BEAQ) was initially simplified and revised by Gámez et al. based on the Multidimensional Experiential Avoidance Questionnaire to assess content related to experiential avoidance. Cao et al. conducted a Chinese version revision in 2021. The questionnaire consists of 15 items, with the cognitive avoidance dimension containing 8 items and the behavioral avoidance dimension containing 7 items, all rated on a 6-point scale from "Strongly Disagree" to "Strongly Agree."
Self-concept | From enrollment to 2 weeks after the completion of the 8-week treatment
  Sense of Mastery Scale, SMS. This scale consists of 12 items, with each item rated on a five-point Likert scale. Higher scores indicate a clearer self-concept among the participants.
meaning in life | From enrollment to 2 weeks after the completion of the 8-week treatment
  The Meaning in Life Questionnaire (MLQ): This scale consists of 10 items with two dimensions: Presence of Meaning (MLQ-P) and Search for Meaning (MLQ-S). Each item adopts a 7-point Likert scale, with higher scores indicating that participants experience a stronger sense of meaning in life.
Grit | From enrollment to 2 weeks after the completion of the 8-week treatment
  The Grit Scale consists of 12 items with two dimensions: the Effort dimension and the Interest Consistency dimension. Each item is rated on a five-point Likert scale, with higher scores indicating that participants perceive themselves as more perseverant.
nature connection | From enrollment to 2 weeks after the completion of the 8-week treatment
  The Nature Connection Scale, which consists of 14 items, employs a 5-point Likert scale for each item, with higher scores indicating that participants perceive themselves as more closely connected to nature.

CONTACTS AND LOCATIONS:
Locations (1):
- Central University of Finance and Economics, Beijing, Beijing 100875, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided